CLINICAL TRIAL: NCT03792880
Title: Global Self-management Telematic Support for Patients With Obstructive Sleep Apnea-hypopnea Syndrome, CPAP Treatment and Forecast of Poor Compliance.
Brief Title: Global Self-management Telematic Support for Patients With Obstructive Sleep Apnea.
Acronym: TELESAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virgen del Puerto Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4/2016
Record Dates: First submitted 2018-10-12; First posted 2019-01-04 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Obstructive Sleep Apnea; Telemedicine; Compliance, Patient
Keywords: CPAP treatment; Self-management
MeSH Terms: conditions — Sleep Apnea, Obstructive; Patient Compliance | interventions — Self-Management; Delivery of Health Care

STUDY DESIGN:
Intervention Model Description: Randomized control trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm (Active Comparator): Usual follow-up in Healthcare System for patients with obstructive sleep apnea and CPAP treatment
  Interventions: Behavioral: Habitual follow-up in Healthcare System
- Intervention arm (Experimental): Usual follow-up in the Healthcare System for patients with obstructive sleep apnea and CPAP treatment and a telematic control and self-management program
  Interventions: Behavioral: Telematic control and self-management program; Behavioral: Habitual follow-up in Healthcare System

INTERVENTIONS:
Behavioral: Telematic control and self-management program — During 6 months with CPAP treatment, patients must complete some questionnaires about the presence of refreshing sleep and side effects with the frequency established, using a computing application. Patients can download this application on their own smartphone but, if they prefer, they can be provided with a tablet during the study with this application installed.
  A set of variables will be collected using an automatic and wireless transmission from latest generation CPAP to control the CPAP compliance and tolerance. All data will be processed in a platform to generate alarms, which will be controled daily by a researcher, as well as solutions to the problems presented during the monitoring.
  Arms: Intervention arm
Behavioral: Habitual follow-up in Healthcare System — According to the SEPAR regulation, patients treated with CPAP should be evaluated by the pulmonologist one month after beginning treatment, every 3 months during the first year, every 6 months during the second year and annually from the third year.

SUMMARY:
This clinical trial compares the usual follow-up to a program of telematic control and self-management in a group of patients with severe obstructive sleep apnea-hypopnea syndrome (OSAHS), few symptoms and treated with continuous positive airway pressure (CPAP). The objective of the intervention is to achieve a CPAP compliance of ≥4 hours per day in at least 90% of the subjects.

DETAILED DESCRIPTION:
Low CPAP compliance in OSAHS could mean that its possible cardiovascular benefits are not achieved. Telemedicine can be an effective tool to increase CPAP compliance with low cost.

The researchers propose to carry out a randomized study about patients with severe OSAHS and few symptoms, who are expected to have low CPAP compliance.

The main objective is to evaluate if a telematic control and self-management program can increase the compliance with CPAP treatment compared to conventional follow-up, getting at least 90% of patients to use CPAP ≥ 4 hours per day.

Sixty patients from the Pneumology departments of two hospitals, diagnosed with severe OSAHS and with few symptoms (Epworth Sleepiness Scale ≤10) will be randomized to two follow-up groups, telematic and conventional, for 6 months. Patients in the intervention group (telematic monitoring) will collect variables related to symptoms of sleep apnea and side effects of CPAP treatment, using their own smartphone or a tablet provided during the study if they prefer. Other variables as the hours per day of CPAP use, leaks and residual apnea-hypopnea index (AHI) will be transmitted daily and automatically from latest generation CPAP. All information will be processed and each variable will generate alarms and instructions for each patient, allowing the self-management and an early solution of the possible problems related to the treatment. Alarms may also be generated in the database if the professional intervention is necessary.

In addition, before starting CPAP treatment and after six months of treatment, patients will be monitored during a week with a watch-like device. Variables related to circadian rhythm will be collected and analyzed to know the effect of CPAP treatment in both groups (control and intervention groups).

ELIGIBILITY:
Inclusion Criteria:

* Patients with a recent diagnostic of OSAHS with AHI≥ 30 and indication of CPAP.
* Age≥ 18 years
* Few symptoms, so that, without hypersomnolence (Epworth sleepiness scale ≤ 10)
* Absence of clinic suspect or confirmation of other sleep pathology
* With interest in the use of new technologies

Exclusion Criteria:

* Nasal obstruction that prevents the use of CPAP
* Psycho-physical inability to complete questionnaires and carry out the program
* Patients undergoing uvulopalatopharyngoplasty
* Cheyne-Stoke syndrome
* Pregnancy
* Absence of informed consent
* Shift work in the last 3 months and transmeridian trips in the last month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-12-28 (Actual); Study Completion 2021-12-28 (Actual)

PRIMARY OUTCOMES:
Patients with a good CPAP compliance | Six months
  Percentage of patients with a CPAP compliance ≥4 hours per day. The main objective is to assess if a self-management and telematic control program can increase CPAP compliance getting at least 90% of patients using CPAP ≥4 hours per day.

SECONDARY OUTCOMES:
CPAP compliance | Six months
  To compare CPAP compliance between both arms using the average compliance (hours of use per day) as secondary variable.
Dropout | Six months
  To compare the dropout percentage between both arms
Side effects | Six months
  To compare the control of side effects between both arms using the percentage of patients who have any of these effects during the follow-up.
Efficacy of the treatment according to the change in sleepiness | Six months
  To compare the efficacy of the treatment using the change of the Epworth Sleepiness Scale score in both arms and between them.
  This scale is a self-administered questionnaire and patients must rate their usual chances of dozing off or falling asleep while engaged in eight different daily activities. The possible answers for each situation and their scores are: 0 = would never doze; 1 = slight chance of dozing; 2 = moderate chance of dozing; 3= high chance of dozing. The Epworth Sleepiness Scale score is the sum of these 8 items scores and it can be interpreted as follows: 0-5 = lower normal daytime sleepiness; 6-10 = higher normal daytime sleepiness; 11-12 = mild excessive daytime sleepiness; 13-15 = moderate excessive daytime sleepiness; 16-24 = severe excessive daytime sleepiness.
Efficacy of the treatment according to the change in the frequency of the snoring. | Six months
  To compare the efficacy of the treatment in both arms and between them using the change in the frequency of the snoring according to four levels: never, sometimes, frequently and always or almost always
Efficacy of the treatment according to the change in the frequency of the witnessed apneas | Six months
  To compare the efficacy of the treatment in both arms and between them using the change in the frequency of the witnessed apneas according to four levels: never, sometimes, frequently and always or almost always
Efficacy of the treatment according to the change in the frequency of the refreshing sleep | Six months
  To compare the efficacy of the treatment in both arms and between them using the change in the frequency of the refreshing sleep according to four levels: never, sometimes, frequently and always or almost always
Presence of air leak and residual AHI | Six months
  To compare the intensity of the air leak and residual AHI measured by the CPAP device between both arms.
Change of quality of life using the change in the EuroQol-5 dimensions-3 levels questionnaire. | Six months
  To compare the change of quality of life before and after the follow-up in both arms and between them, using the change in the EuroQol-5 dimensions-3 levels questionnaire. This is a standardised measure of health status that comprises a descriptive system and a visual analogue scale. The first comprises 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: 1 = no problems; 2 = some or moderate problems; 3 = extreme problems. The health state is defined by combining one level from each dimension (5 digit code). This descriptive system is converted into a single index value facilitating comparisons and the calculation of quality-adjusted life years (QALYs). The visual analogue scale records the respondent's self-rated health on a 20 centimeters vertical, visual analogue scale with endpoints labeled as: 100 = the best health you can imagine and 0. = the worst health you can imagine.
Effect of the treatment in the quality of sleep using the change in the rhythm of the distal skin temperature. | Six months
  To compare the effect of the treatment in the quality of sleep using the change in the rhythm of distal skin temperature by ambulatory circadian monitoring including this variable. The investigators will compare the rhythm of this variable before and after CPAP treatment in both arms and the difference between them. For this propose, all randomized patients will carry a watch-like device for ambulatory circadian monitoring during one week before starting CPAP treatment and during the last week of the six months of follow-up and treatment with CPAP.
Effect of the treatment in the quality of sleep using the change in the rhythm of activity. | Six months
  To compare the effect of the treatment in the quality of sleep using the change in the rhythm of activity by ambulatory circadian monitoring including this variable. The investigators will compare the rhythm of this variable before and after CPAP treatment in both arms and the difference between them. For this propose, all randomized patients will carry a watch-like device for ambulatory circadian monitoring during one week before starting CPAP treatment and during the last week of the six months of follow-up and treatment with CPAP.
Effect of the treatment in the quality of sleep using the change in the rhythm of exposure to light | Six months
  To compare the effect of the treatment in the quality of sleep using the change in the rhythm of exposure to light by ambulatory circadian monitoring including this variable. The investigators will compare the rhythm of this variable before and after CPAP treatment in both arms and the difference between them. For this propose, all randomized patients will carry a watch-like device for ambulatory circadian monitoring during one week before starting CPAP treatment and during the last week of the six months of follow-up and treatment with CPAP.
Effect of the treatment in the quality of sleep using the change in the result of an integrated analysis of the distal skin temperature, activity and position records. | Six months
  To compare the effect of the treatment in the quality of sleep using the change in the result of an integrated analysis of the distal skin temperature, activity and position records obtained by ambulatory circadian monitoring including these variables. The researchers will compare this result before and after CPAP treatment in both arms and the difference between them. For this propose, all randomized patients will carry a watch-like device for ambulatory circadian monitoring during one week before starting CPAP treatment and during the last week of the six months of follow-up and treatment with CPAP.
Effect of the presence of a couple on the treatment efficacy. | Six months
  To compare the efficacy of the treatment according to the presence or not of a couple, comparing the percentage of patients with CPAP compliance ≥4 hours per day between both groups of patients (all patients with and without couple), within each arm (control and intervention arm) and between arms.
Effect of the age on the treatment efficacy | Six months
  To analyze the influence of the patients' age on the percentage of patients with a CPAP compliance ≥4 hours per day in both arms.
Effect of the gender on the treatment efficacy | Six months
  To compare the efficacy of the treatment depending on the gender, comparing the percentage of patients with a CPAP compliance ≥4 hours per day between all men and all women, within each arm and between arms.
Effect of the CPAP pressure on the treatment efficacy | Six months
  To analyze the effect of the CPAP pressure on the percentage of patients with a CPAP compliance ≥4 hours per day in both arms.
Effect of the type of mask on the treatment efficacy | Six months
  To compare the efficacy of the treatment depending on the type of mask used during the CPAP treatment, comparing the percentage of patients with a CPAP compliance ≥4 hours per day in the group of patients who use nasal pillow, full face and nasal mask in both arms and between them.
Effect of the use of humidifier on the treatment efficacy | Six months
  To compare the efficacy of the treatment depending on the use of humidifier during the CPAP treatment, comparing the percentage of patients with a CPAP compliance ≥4 hours per day in the group of patients who use or not humidifier in both arms and between them.
Effect of the presence of side effects on the treatment efficacy | Six months
  To compare the efficacy of the treatment depending on the presence of any side effect during the CPAP treatment, comparing the percentage of patients with a CPAP compliance ≥4 hours per day in the group of patients with and without any side effect in both arms and between them.
Cost-effectiveness analysis | Six months
  The researchers will perform a cost-effectiveness analysis using the average compliance as main variable of effectiveness, and the EuroQol-5 dimensions-3 levels descriptive system to calculate QALYs.
  EuroQol-5 dimensions-3 levels descriptive system is a standardised measure of health status that comprises 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: 1 = no problems; 2 = some or moderate problems; 3 = extreme problems. The respondent have to indicate his/her health state according to the most appropiate statement in each dimension. The health state is defined by combining one level from each of the 5 dimensions (5 digit code) and then, this descriptive system is converted into a single index value facilitating comparisons and the calculation of quality-adjusted life years (QALYs).

CONTACTS AND LOCATIONS:
Overall Officials: María Ángeles Sánchez Quiroga, Principal Investigator — Virgen del Puerto Hospital
Locations (2):
- Spain (2):
  - Virgen del Puerto Hospital, Plasencia, Cáceres
  - San Pedro de Alcántara, Cáceres